CLINICAL TRIAL: NCT03675243
Title: Quality of Life After Transanal Endoscopic Microsurgery (TEM) for Rectal Neoplasm
Brief Title: Quality of Life After Transanal Endoscopic Microsurgery (TEM)
Acronym: QoLTEM
Status: Completed | Type: Observational
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Sponsor
Other Study IDs: 85A
Record Dates: First submitted 2018-09-12; First posted 2018-09-18 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Transanal Endoscopic Microsurgery (TEM)
Keywords: Transanal endoscopic microsurgery; TEM; QoL; quality of life; rectal cancer; rectal surgery; rectal neoplasm
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: sphincterometry — Sphincterometry is a method of the spincter function examination, which allows to assess the state of the anal sphincter muscle and its function

SUMMARY:
This is a observational cohort study to determine the influence of Transanal endoscopic microsurgery (TEM) on patients Quality of Life

DETAILED DESCRIPTION:
Patients who planning Transanal Endoscopic Microsurgery (TEM) for rectal neoplasms should undergoing fecal incontinence quality of life scale and Wexner score before and after surgery for measurement their quality of life. For objectification data sphinctrometry will be perform.

ELIGIBILITY:
Inclusion Criteria:

* Have a planned of Transanal endoscopic microsurgery (TEM)
* Have signed approved informed consent form for the study

Exclusion Criteria:

* non epithelial malignancy
* recurrent neoplasm
* stoma formation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rectal neoplasms with planning transanal endoscopic microsurgery (TEM)
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Fecal incontinence quality of life scale | 3 month
  The FIQL is a standardized instrument that can be used to assess QOL issues related to fecal incontinence.The Fecal Incontinence Quality of Life Scale is composed of a total of 29 items; these items form four scales: Lifestyle (10 items), Coping/Behavior (9 items), Depression/Self-Perception (7 items), and Embarrassment (3 items).Each aspect is described as a score measured on a scale between 1 and 4, where 1 is very affected and 4 is not affected

SECONDARY OUTCOMES:
Wexner score | 3 month
  Wexner score is composed of a total 5 items for each type of incontinence. Each aspect is described as a score measured on a scale between 1 and 4, where 0 is rarely, 4 - always/ 0 - perfect, 20 - complete incontinence.
Sphinctrometry | 3 month
  Anal pressure in mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- State Scientific Centre of Coloproctology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No